CLINICAL TRIAL: NCT02037035
Title: Examining The Effect Of Ketamine On Glutamate/Glutamine Cycling
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); American Psychiatric Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1305011972; 1K23MH101498-01 (NIH)
Record Dates: First submitted 2013-11-19; First posted 2014-01-15 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy (Experimental): Healthy participants will receive ketamine in the scan
  Interventions: Drug: Ketamine
- Depressed (Experimental): Depressed participants will receive ketamine in the scan
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine

SUMMARY:
This study is looking at the mechanisms underlying the behavioral effects of ketamine in healthy and depressed individuals.

ELIGIBILITY:
Healthy Group

Inclusion Criteria:

* Male or female between the ages of 21-65 years.
* Able to provide written informed consent.
* Able to read and write English.

Exclusion Criteria:

* Personal or first-degree family member with history of mood, anxiety, or psychotic axis I DSM-IV disorders confirmed after comprehensive psychiatric evaluation.
* Any history of serious medical or neurological illness.
* Any signs of major medical or neurological illness on examination or as a result of ECG screening or laboratory studies.
* Lifetime history of psychoactive substance or alcohol dependence or substance or alcohol abuse (other than nicotine or caffeine abuse), or drinking more that 5 drinks/week during the last year.
* Abnormality on physical examination.
* A positive pre-study (screening) urine drug screen or, at the study physician's discretion on any drug screens given before the scans.
* Pregnant or lactating women or a positive urine pregnancy test for women of child-bearing potential at screening or prior to any imaging day.
* Subjects who test positive for HIV or viral hepatitis (hepatitis B and/or C)
* Has received either prescribed or over-the-counter (OTC) centrally active medicine or herbal supplements within the week prior to the MRI scan.
* Any history indicating learning disability, mental retardation, or attention deficit disorder.
* Known sensitivity to ketamine.
* Body circumference of 52 inches or greater.
* Body weight of 280 pounds or greater.
* History of claustrophobia.
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI screening questionnaire.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Resting blood pressure lower than 90/60 or higher than 150/90,or resting heart rate lower than 45/min or higher than 100/min.

Depression Group

Inclusion Criteria:

* Male or female between the ages of 21-65 years.
* Able to provide written informed consent.
* Current MDD Single Episode (296.2x) or Recurrent (296.3x), as determined by the Structured Clinical Interview for DSM-IV (SCID) patient edition
* Montgomery Asberg Depression Rating Scale (MADRS) score of 18 or higher at baseline and start of first 13C-MRS.
* Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR16) score of 19 or higher at baseline and start of first 13C-MRS.
* No psychotropic medications for 2 or more weeks (4 weeks for Fluoxetine) prior to first 13C-MRS.
* Be able to understand and speak English.

Exclusion Criteria:

* Patients with a history of DSM-IV-TR diagnosis of bipolar disorder or schizophrenia or schizoaffective disorder or currently exhibiting psychotic features associated with their depression; dementia or suspicion thereof, is also exclusionary.
* First-degree family member with history of schizophrenia or any other psychotic disorder.
* Serious suicide or homicide risk, as assessed by evaluating clinician; A serious suicide risk will be considered an inability to control suicide attempts, imminent risk of suicide in the investigator's judgment, or a history of serious suicidal behavior, which is defined using the Columbia-Suicide Severity Rating Scale (C-SSRS) as either (1) one or more actual suicide attempts in the 3 years before study entry with the lethality rated at 3 or higher, or (2) one or more interrupted suicide attempts with a potential lethality judged to result in serious injury or death.
* Substance abuse or dependence during the 12 months prior to screening.
* Any history of serious medical or neurological illness.
* Any signs of major medical or neurological illness.
* Abnormality on physical examination. A subject with a clinical abnormality may be included only if the study physician considers the abnormality will not introduce additional risk factors and will not interfere with the study procedure.
* A positive pre-study (screening) urine drug screen or on any drug screens given before the scans.
* Pregnant or lactating women or a positive urine pregnancy test for women of childbearing potential at screening or prior to any imaging day.
* Any history indicating learning disability, or mental retardation.
* Known sensitivity to ketamine.
* Body weight of 280 pounds or greater.
* History of claustrophobia.
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI screening questionnaire.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Resting blood pressure lower than 90/60 or higher than 150/90,or resting heart rate lower than 45/min or higher than 100/min.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Glutamate Metabolism | 40-75 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette Averill, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Depression Research Program, New Haven, Connecticut, United States